CLINICAL TRIAL: NCT00176475
Title: A Pilot Study of Irradiated HLA-Partially Matched Allogeneic Related Donor Lymphocytes in Conjunction With Rituximab for Selected Patients With CD20 + Malignancies
Brief Title: Irradiated Donor Lymphocytes and Rituximab in Treating Patients With Relapsed or Refractory Lymphoproliferative Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000540171; P30CA072720 (NIH); CINJ-010406 (Other: Cancer Institute of New Jersey)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; recurrent small lymphocytic lymphoma; refractory hairy cell leukemia; prolymphocytic leukemia; recurrent marginal zone lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; refractory multiple myeloma; recurrent mantle cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; Waldenstrom macroglobulinemia; splenic marginal zone lymphoma; stage II multiple myeloma; stage III multiple myeloma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; progressive hairy cell leukemia, initial treatment
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Prolymphocytic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic allogeneic lymphocytes with rituximab (Experimental)
  Interventions: Biological: rituximab; Biological: therapeutic allogeneic lymphocytes

INTERVENTIONS:
Biological: rituximab — Patients will receive a single day infusion of standard dose rituximab (375 mg/m2) on days -1, 6, 13, 20 approximately every 4 months (in conjunction with alternating doses of the lymphocyte infusion).
Biological: therapeutic allogeneic lymphocytes — The product will then be assigned to the specific patient and the released product will be transported to and administered to the patient at CINJ, after premedication of the patient with acetaminophen 650 mg PO and diphenhydramine- HCl 25 mg PO. Blood product administration will be every 8 weeks and undertaken according to CINJ standard procedures

SUMMARY:
RATIONALE: When irradiated lymphocytes from a donor are infused into the patient they may help the patient's immune system kill cancer cells. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving irradiated donor lymphocytes together with rituximab may kill more cancer cells.

PURPOSE: This clinical trial is studying the side effects and how well giving irradiated donor lymphocytes together with rituximab works in treating patients with relapsed or refractory lymphoproliferative disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity of irradiated HLA-partially matched related donor lymphocytes when administered with rituximab in patients with relapsed or refractory CD20-positive lymphoproliferative disease.
* Determine the efficacy of this regimen in these patients.

Secondary

* Correlate response with Fc receptor FcγIIIA polymorphisms or predicted HLA-directed natural killer cell reactivity.

OUTLINE: This is a pilot study.

* Rituximab therapy: Patients receive rituximab IV on days -1, 6, 13, and 20. Treatment repeats approximately every 4 months in the absence of disease progression or unacceptable toxicity.
* Donor lymphocyte infusion: Patients receive irradiated donor lymphocytes IV over 1 hour on day 0. Treatment repeats every 8-16 weeks (alternating with courses of rituximab therapy) for up to 6 donor lymphocyte infusions in the absence of disease progression or unacceptable toxicity.

Peripheral blood is collected periodically during study for correlative laboratory studies. Blood samples are analyzed for FcγIIIA polymorphism by fluorescent in situ hybridization or by reverse transcriptase-polymerase chain reaction. Survival of donor lymphocytes is assessed by chimerism studies.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed lymphoproliferative disease

  * CD20-positive disease
* Bidimensionally measurable disease OR abnormal cells detected in blood
* Resistant or refractory to standard therapies and/or unlikely to benefit from additional standard therapies* AND meets 1 of the following criteria:

  * Disease with anticipated response rate < 20% after treatment with rituximab alone, including any of the following:

    * Diffuse large cell lymphoma
    * B-cell lymphoblastic lymphoma
    * Burkitt's lymphoma
    * Acute lymphocytic leukemia
  * Relapsed or progressive disease after prior treatment with rituximab, including any of the following:

    * Hodgkin's lymphoma
    * Hairy cell leukemia
    * Chronic lymphocytic leukemia/small lymphocytic lymphoma meeting any of the following criteria:

      * Received prior fludarabine phosphate-containing regimens and relapsed within 1 year of treatment OR ineligible to receive such therapy due to comorbidities or allergies
      * Received prior anti-CD52 monoclonal antibody therapy and relapsed within 1 year of treatment OR ineligible to receive such therapy (for patients without symptomatic lymphadenopathy)
      * Has documentation of disease-associated symptoms, rapid disease progression, or other indications for treatment
    * B-cell prolymphocytic leukemia meeting any of the following criteria:

      * Received prior fludarabine phosphate- or alkylating agent-containing regimens and relapsed within 1 year of treatment OR ineligible to receive such therapy due to comorbidities or allergies
      * Received prior anti-CD52 monoclonal antibody therapy OR ineligible to receive such therapy (for patients without symptomatic lymphadenopathy)
    * Lymphoplasmacytic lymphoma, marginal zone lymphoma, mucosa-associated lymphoid tissue lymphoma, or follicular lymphoma meeting any of the following criteria:

      * Received prior fludarabine phosphate- and/or alkylating agent-containing regimens and relapsed within 1 year of treatment OR ineligible to receive such therapy due to comorbidities or allergies
      * Received prior anti-CD20 monoclonal antibody therapy and relapsed within 1 year of treatment OR ineligible to receive such therapy
      * Received prior radioconjugated anti-CD20 monoclonal antibody therapy OR ineligible to receive such therapy
      * Has documentation of disease-associated symptoms, rapid disease progression, or other indications for treatment
    * Multiple myeloma meeting any of the following criteria:

      * Received prior alkylating agent-, thalidomide-, corticosteroid-, or bortezomib-containing regimens and relapsed after 1 year of treatment OR ineligible to receive such therapies due to comorbidities or allergies
      * Received prior high-dose chemotherapy followed by autologous hematopoietic stem cell rescue and relapsed after treatment OR ineligible to receive such therapy
    * Mantle cell lymphoma meeting the following criteria:

      * Received prior combination chemotherapy and anti-CD20 monoclonal antibody therapy and relapsed after treatment OR ineligible to receive such therapy
    * Diffuse large B-cell lymphoma meeting any of the following criteria:

      * Received prior combination chemotherapy and relapsed after treatment OR ineligible to receive such therapy
      * Received prior salvage combination chemotherapy with or without high-dose chemotherapy followed by autologous hematopoietic stem cell rescue and relapsed after treatment OR not a candidate to receive such therapy
      * Received prior radiolabeled anti-CD20 monoclonal antibody therapy for transformed large cell lymphoma OR ineligible to receive such therapy
    * Burkitt's lymphoma meeting any of the following criteria:

      * Received prior combination chemotherapy and relapsed after treatment OR ineligible to receive such therapy
      * Received prior salvage combination chemotherapy with or without high-dose chemotherapy followed by autologous hematopoietic stem cell rescue and relapsed after treatment OR ineligible to receive such therapy
    * Lymphomatoid granulomatosis meeting any of the following criteria:

      * Received prior single-agent or combination chemotherapy and relapsed after treatment OR ineligible to receive such therapy
      * Has documentation of disease-associated symptoms, rapid disease progression, or other indications for treatment
    * Acute lymphocytic leukemia meeting any of the following criteria:

      * Received prior multi-agent combination chemotherapy administered in sequential induction, consolidation, and maintenance courses and relapsed during or after treatment OR ineligible to receive such therapy
      * Received prior chemotherapy with or without radiotherapy followed by allogeneic hematopoietic stem cell transplantation (HSCT) and relapsed after treatment OR not a candidate for such therapy
      * Received prior treatment with chemotherapy with or without radiotherapy followed by allogeneic HSCT and relapsed after treatment (or not a candidate for such therapy) AND demonstrates persistent cytogenetic, fluorescent in situ hybridization, or molecular (reverse transcriptase-polymerase chain reaction) evidence of the bcr-abl fusion gene despite 6 weeks of treatment with imatinib mesylate NOTE: *Not eligible to receive standard available salvage regimens anticipated to result in durable remission
* No active CNS malignancy
* Not considered a candidate for allogeneic HSCT
* HLA-partially matched (≥ 2/6) related donor available

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 3 months
* Not pregnant
* Negative pregnancy test
* Fertile women must use effective contraception
* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST < 3.0 times ULN
* Cardiac ejection fraction > 35%
* Absolute neutrophil count > 1,000/mm³ (without cytokines)
* Platelet count > 50,000/mm³ (untransfused)
* No significant organ dysfunction
* No active uncontrolled infections
* No hypersensitivity reaction to rituximab that has precluded completion of a 4-week course of rituximab therapy
* No uncontrolled psychiatric illness or medical condition that would preclude tolerance of study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy for at least 7 days
* More than 30 days since prior cytotoxic chemotherapy
* At least 14 days since prior steroids
* At least 14 days since prior radiotherapy to non-target lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Toxicity as assessed by NCI CTCAE v3.0 | 4 years

SECONDARY OUTCOMES:
Efficacy | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States